CLINICAL TRIAL: NCT04178148
Title: Personalized Dose Optimization of Amikacin Guided by Pharmacokinetic Modeling Software in Patients With Septic Shock
Acronym: AMINO BESTDOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2018-02/CR-01
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Shock, Septic
Keywords: Pharmacokinetics; dose optimisation; aminoglycosides
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BestDose (Experimental): Therapeutic drug optimization of amikacin using the BestDose software algorithm
  Interventions: Other: Amikacin dose optimization
- Control (No Intervention)

INTERVENTIONS:
Other: Amikacin dose optimization — Therapeutic drug optimization of amikacin using the BestDose software algorithm
  Arms: BestDose

SUMMARY:
Amikacin dose optimization is challenging in critically ill patients. The use of BestDose software algorithm-based drug optimization could help to achieve the recommended target concentrations (60-80 mg/L) after administration of the second dose of amikacin, associated with improved outcome. The study investigators hypothesize that 80% of patients undergoing drug dosing optimization using the BestDose software in the interventional group will reach the predefined PK/PD targets.

ELIGIBILITY:
Inclusion Criteria:

* The patient or their legal representative must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient has septic shock according to the SEPSIS-3 definition in the 24 hours preceding inclusion, regardless of the source of infection
* Patient having already received a first dose of amikacin in the 22 preceding hours
* Patient with an expectation of receiving at least 2 doses of amikacin
* Patient with available amikacin therapeutic drug monitoring

Exclusion Criteria:

* The subject is participating in an interventional study that could influence the primary outcome, or is in a period of exclusion determined by a previous study
* The patient is pregnant, parturient or breastfeeding
* Patient has a contra-indication or an allergy to treatment by amikacin
* Patient is not expected to survive beyond 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Patients reaching target amikacin maximum concentration following second dose | 30 minutes after second dose of amikacin
  Yes/no; Cmax 60-80mg/l

SECONDARY OUTCOMES:
Patients reaching target amikacin minimum concentration following second dose | 24 hours after second dose of amikacin
  Yes/no
Patients reaching target amikacin maximum concentration following third dose | 30 minutes after third dose of amikacin
  Yes/no; Cmax 60-80mg/l
Patients reaching target amikacin minimum concentration following third dose | 24 hours after third dose of amikacin
  Yes/no
Time taken to reach recommended Cmax during amikacin therapy | Maximum 7 days
  Hours
Clinical cure test | At end of treatment (Maximum day 7)
  Either clinical-evaluated or assessed according to patient medical files: classified as resolved, improved, failed
Clinical cure test | Day 7
  Either clinical-evaluated or assessed according to patient medical files: classified as resolved, improved, failed
Number of days without renal replacement therapy | Day 28
  Number
Number of days without vasopressors | Day 28
  Number
Number of days without mechanical ventilation | Day 28
  Number
Mortality | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roger, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

REFERENCES:
- [Result] Garbez N, Mbatchi LC, Louart G, Wallis SC, Muller L, Lipman J, Roberts JA, Lefrant JY, Roger C. Micafungin Population PK Analysis in Healthy and Septic Pigs: Can the Septic Porcine Model Predict the Micafungin PK in Septic Patients? Pharm Res. 2021 Nov;38(11):1863-1871. doi: 10.1007/s11095-021-03137-2. Epub 2021 Nov 29. PMID 34845574